CLINICAL TRIAL: NCT05210933
Title: Study of Minimally-invasive Ablative Renal Therapies (SMART) Registry
Acronym: SMART
Status: Suspended | Type: Observational
Why Stopped: Study is currently on hold.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: HREBA.CC-20-0432
Record Dates: First submitted 2021-12-13; First posted 2022-01-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Renal Cancer
Keywords: renal cancer; cryoablation; small renal mass
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood and urine samples will be collected at baseline (i.e. study entry), and once after treatment is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multi-center prospective cohort study examining curative intent renal cryotherapy and radiofrequency ablation for small renal mass treatment in patients who are poor candidates for surgical resection, We will capture clinical, radiological, and pathological data as well as resource utilization (ex: time in hospital, ER visits), complications, and long-term functional and oncological outcomes. The investigators will also be biobanking blood and urine samples from participants for biological studies in the lab.

DETAILED DESCRIPTION:
Currently the standard-of-care for non-operative renal masses which require treatment is curative ablative therapy. Curative ablative therapies include radiofrequency ablation (RFA) and cryotherapy. A significant number of patients (approximately 40-50%) can only be treated with cryotherapy rather than RFA because of the target lesions close proximity to the collecting system, ureter, solid organs or hollow viscera. Cryotherapy allows for size control of the ablation zone with CT surveillance to avoid iatrogenic injury to these vital structures. On the other hand RFA does not allow for the same ability to control the size of ablation and, unfortunately due to the thermal energy, can result in injury to these structure precluding the use of RFA as a curative therapy for these patients.

Cryoablation of small renal masses provides equivalent intermediate-term cancer control compared to partial nephrectomy. Three-year local recurrence-free survival is 98% for both cryoablation and partial nephrectomy. Similarly metastasis-free survival three years after treatment is 100% for cryoablation and 99% for partial nephrectomy. Curative renal mass ablations provide the added benefit of being outpatient procedures which do not routinely require more than a 4 hour post-procedural recovery and over-the-counter post-procedural analgesic.

Research Question and Objectives:

The objective is to to provide cryotherapy and RFA as curative treatment options for small renal mass treatment in patients who are poor candidates for surgical resection or for those who are not surgical candidates due to co-morbidities. The investigators aim to establish a database that prospectively captures clinical, radiological, and pathological data as well as resource utilization (ex: time in hospital, ER visits), complications, and long-term functional and oncological outcomes. The study will also be biobanking blood and urine samples from participants for biological studies in the lab.

Methods:

Program Design Ablation to be performed percutaneously under CT/ultrasound guidance at the Royal Alexandra Hospital in Edmonton or the Rocky View Health Centre in Calgary, by a team of Interventional Radiologists and Urologists. A CT technologist, Ultrasound technologist and an Interventional Radiologist/Urologist are required for each procedure.

Each patient must have cross sectional imaging (CT or MRI) to confirm that they are a candidate to be treated with curative ablative therapy and to plan the procedure.

Pre-procedural consults by both the Urologist and IR performing the procedure. Patients to be assessed in the diagnostic imaging recovery room (DIRR) prior to the procedure and post-procedure to return to the DIRR or OR recovery room. Procedure to be performed with anesthesia support for deep sedation. Post treatment follow-up will be in accordance with the Canadian Urological Associations published guidelines

Blood and urine samples will be collected at baseline (i.e. study entry), yearly during follow-up for 5 years, and when changes occur in cancer status, for example after radical kidney therapy (surgical removal) or after disease progression (new metastases) during the study's potential observation period.

In addition to the samples, an intake survey must be completed at baseline and ongoing questionnaires completed by participant once a year for five years and when new cancer problems arise until up to five years.

ELIGIBILITY:
Inclusion Criteria:

* Adults with prior kidney tumor diagnosis;
* Willing to permit provincial agencies (e.g Alberta Health Services, Alberta Health, Netcare, Service Alberta) to disclose health-related information to study;
* Canadian and Albertan residents;
* Signed informed consent.

Exclusion Criteria:

* Unwilling to participate in the study;
* Unavailable for standard clinical urological care or follow-up in Alberta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Albertans with a diagnosis of kidney cancer
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
kidney cancer disease-specific survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival will be calculated in years (Mean and Median will be calculated)
Glomerular Filtration Rate GFR (mL/min/1.73m2) | 5 years
  Renal function measured in Glomerular Filtration Rate GFR (mL/min/1.73m2)
Serum Creatinine (umol/L) | 5 years
  Renal function measured in Serum Creatinine (umol/L). Serum Cr will be collected pre-cryotherapy and every 3-6 months following for five years as per Canadian Urological Association Guidelines and our study protocol.
Progression-free survival | 5 years
  Local and metastatic disease recurrence measured in years

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

REFERENCES:
- [Background] Kassouf W, Monteiro LL, Drachenberg DE, Fairey AS, Finelli A, Kapoor A, Lattouf JB, Leveridge MJ, Power NE, Pouliot F, Rendon RA, Sabbagh R, So AI, Tanguay S, Breau RH. Canadian Urological Association guideline for followup of patients after treatment of non-metastatic renal cell carcinoma. Can Urol Assoc J. 2018 Aug;12(8):231-238. doi: 10.5489/cuaj.5462. Epub 2018 May 31. No abstract available. PMID 30139427
- [Background] Thompson RH, Atwell T, Schmit G, Lohse CM, Kurup AN, Weisbrod A, Psutka SP, Stewart SB, Callstrom MR, Cheville JC, Boorjian SA, Leibovich BC. Comparison of partial nephrectomy and percutaneous ablation for cT1 renal masses. Eur Urol. 2015 Feb;67(2):252-9. doi: 10.1016/j.eururo.2014.07.021. Epub 2014 Aug 6. PMID 25108580